CLINICAL TRIAL: NCT01525875
Title: Magnesium Supplements In The Treatment Of Pseudoxanthoma Elasticum (PXE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mark Lebwohl (Other)
Responsible Party: Sponsor-Investigator, Mark Lebwohl, Principal Investigator, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GCO 09-1157; FD-R-0003903 (Other Grant/Funding Number: FDA OOPD)
Record Dates: First submitted 2012-02-01; First posted 2012-02-03 (Estimated); Results first posted 2019-04-25 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-02

CONDITIONS: Pseudoxanthoma Elasticum
Keywords: pseudoxanthoma elasticum; calcification
MeSH Terms: conditions — Pseudoxanthoma Elasticum; Calcinosis | interventions — Magnesium Oxide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Magnesium oxide (Active Comparator): Part 1: 1000 mg elemental magnesium (given as one 800 mg capsule of magnesium oxide two times daily).
  Part 2: 1500 mg elemental magnesium (given as two 500 mg capsules of magnesium oxide in the morning and three 500 mg capsules of magnesium oxide in the evening).
  Interventions: Drug: Magnesium Oxide
- Placebo (Placebo Comparator): Part 1: 1000 mg (one 500 mg capsule two times daily) of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Magnesium Oxide — Part 1: 1000 mg elemental magnesium (given as one 800 mg capsule of magnesium oxide two times daily).
  Part 2: 1500 mg elemental magnesium (given as two 500 mg capsules of magnesium oxide in the morning and three 500 mg capsules of magnesium oxide in the evening).
  Other Names: magnesium oxide supplement
  Arms: Magnesium oxide
Drug: Placebo — 1000 mg (one 500 mg capsule two times daily) of placebo.
  Other Names: silica and/or cellulose
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effectiveness of magnesium oxide supplements on the reversal of calcium deposits in the skin, and the yellow bumps and folds of skin in subjects with pseudoxanthoma elasticum (PXE). Magnesium oxide is a dietary supplement that has been shown in some research to reduce these calcium deposits. This study consists of two parts. The first part is a year-long, double-blind, placebo-controlled study. Part two is an open-label, year-long study. In Part 1, qualified subjects will be randomized to receive either magnesium oxide supplements or placebo, in a 1:1 ratio for the first 12 months. The starting dose will be 1000 mg daily, and depending on tolerability, doses may be decreased. Baseline evaluations will be comprised of: blood tests; clinical evaluations; skin biopsy; eye examination; bone density test; and photography of skin lesions. Subjects will be evaluated at week 2, week 6, month 3, and then every 3 months during the first year. Upon completion of the first year, barring any safety concerns, all subjects will be administered magnesium oxide supplements for up to one additional year. Subjects will undergo the same evaluations/ procedures every 3 months. We hypothesize that the magnesium oxide will cause a reduction in calcifications in the subject's soft tissue/skin. Funding Source - FDA OOPD.

DETAILED DESCRIPTION:
Pseudoxanthoma elasticum (PXE) is a systemic connective tissue disorder involving elastic fiber calcification and fragmentation with major clinical manifestations occurring in the cutaneous, ocular and cardiovascular systems.

Calcification of the elastic fibers leads to cracks in Bruch's membrane, an elastic tissue-containing membrane that separates the vascular choroid from the retinal pigment epithelium. These are known as angioid streaks and may be the only sign of the disease for years. Retinal hemorrhage and loss of vision are common. Calcification of the internal elastic lamina of arteries results in gastrointestinal bleeding, sometimes fatal in nature. Accelerated heart disease is an additional complication.

Cutaneous manifestations are characterized by the presence of yellow papules in a cobblestone pattern or plaques resembling "plucked chicken-skin" in flexural regions. Redundant folds of skin may develop in more advanced cases. The most frequent sites of cutaneous involvement include the neck, axillae, inguinal region, antecubital and popliteal fossae and the periumbilical area. Skin lesions provide an easy way of grading degree of calcification of elastic tissue.

A clinical study of 80 subjects with a variety of cutaneous soft tissue mineralization disorders had the affected areas injected locally with magnesium sulfate while also receiving oral magnesium lactate for 4 to 6 months. About 75% of these subjects showed a significant decrease or complete disappearance of calcification.

More recently, a knockout mouse model for PXE has linked a reversal in calcification to a diet high in magnesium. Mice were placed on diets that were either high or low in phosphate, high or low in magnesium, or on a controlled diet. The mice placed on the high magnesium diet did not show any evidence of connective tissue mineralization, while those on the other diets did show mineralization as characterized by calcification of the connective tissue capsule surrounding the vibrissae.

Based on this information and the research linking increased magnesium levels to decreased calcification, we plan to supplement the diets of PXE patients with magnesium oxide in order to show a reduction in elastic fiber calcification in the skin and to slow the progression of the disease.

Randomized subjects will be instructed to take study drug (active or placebo) for 12 months, then all subjects will receive active study drug for the following 12 months.

When ingested through foods, magnesium has not demonstrated any adverse effects. When obtained through supplements, however, excessive magnesium intake has been known to result in diarrhea as well as other gastrointestinal effects such as nausea, and abdominal cramping. Large pharmacological doses of magnesium have been associated with more serious side effects, such as metabolic alkalosis and hypokalemia with the repeated daily ingestion of 30g of magnesium oxide. Hypermagnesemia may result with excessive magnesium supplement ingestion, however, it has rarely been reported in individuals with normal renal function.

Study data will be analyzed using the Wilcoxon Rank Sum Test to compare changes in physician global assessment of skin lesions, evaluation of target lesions and assessment of biopsies between treatment and placebo groups. Assuming a negligible placebo response, we believe power analyses can be performed on our primary measure in 40 completed subjects as proposed in this study. Analyses will be based on intent-to-treat, with the last observation carried forward. Patients who withdraw for safety, lack of efficacy, and generally those without other documentation will in the absence of the requested 'final-visit evaluation' be assigned the highest (worst) score. A finding of significance based on the intent-to-treat analysis would be supplemented with an analysis of patients completing the trial without any protocol deviations.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject at least 18 years of age
* If female, the subject is not pregnant or nursing
* If female of child bearing potential, the subject has a negative urine pregnancy test at the first visit, and agrees to use an approved method of contraception (hormonal contraceptives [birth control pills, implants [Norplant] or injections [DepoProvera]); intrauterine device (IUD); two forms of barrier methods [condoms and diaphragm]; or abstinence (no sexual activity) throughout the entire study
* Biopsy confirmed diagnosis of pseudoxanthoma elasticum (documenting some calcification of elastic fibers)
* Subject has a clinical disease severity grade of at least "1" (Poorly defined, barely visible macules) at screening.
* Normal kidney function tests

Exclusion Criteria:

* Any subject who is pregnant or becomes pregnant during the study
* Subjects with a serum creatinine greater than 1.6 mg/dL
* Subjects with hypermagnesemia, hypokalemia, or idiopathic hypercalciuria
* Subjects with kidney disease or renal tubular defects (eg. Fanconi's syndrome), or on dialysis
* Subjects with hypothyroidism or hypoparathyroidism or primary hyperparathyroidism
* Subjects with acute gout
* Subjects with malabsorption, or osteomalacia
* Subjects on diuretics, magnesium containing antacids, or anabolic steroids
* Subjects with Cushing's syndrome
* Subjects receiving lithium and those with significant psychiatric disorders that would likely interfere with participation in this study
* Subjects taking anti-seizures medications and anti-arrhythmics medications
* Subjects on tetracycline or metronidazole and ace inhibitors
* Subjects taking cyclosporine or calcineurin inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-08; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Lebwohl, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lebwohl M, Neldner K, Pope FM, De Paepe A, Christiano AM, Boyd CD, Uitto J, McKusick VA. Classification of pseudoxanthoma elasticum: report of a consensus conference. J Am Acad Dermatol. 1994 Jan;30(1):103-7. doi: 10.1016/s0190-9622(08)81894-4. No abstract available. PMID 8277008
- [Background] Neldner KH. Pseudoxanthoma elasticum. Clin Dermatol. 1988 Jan-Mar;6(1):1-159. doi: 10.1016/0738-081x(88)90003-x. No abstract available. PMID 3359381
- [Background] Clarkson JG, Altman RD. Angioid streaks. Surv Ophthalmol. 1982 Mar-Apr;26(5):235-46. doi: 10.1016/0039-6257(82)90158-8. PMID 7046115
- [Background] Renie WA, Pyeritz RE, Combs J, Fine SL. Pseudoxanthoma elasticum: high calcium intake in early life correlates with severity. Am J Med Genet. 1984 Oct;19(2):235-44. doi: 10.1002/ajmg.1320190205. PMID 6507474
- [Background] Martinez-Hernandez A, Huffer WE, Neldner K, Gordon S, Reeve EB. Resolution and repair of elastic tissue calcification in pseudoxanthoma elasticum. Arch Pathol Lab Med. 1978 Jun;102(6):303-5. PMID 580723
- [Background] Sapadin AN, Lebwohl MG, Teich SA, Phelps RG, DiCostanzo D, Cohen SR. Periumbilical pseudoxanthoma elasticum associated with chronic renal failure and angioid streaks--apparent regression with hemodialysis. J Am Acad Dermatol. 1998 Aug;39(2 Pt 2):338-44. doi: 10.1016/s0190-9622(98)70385-8. PMID 9703148
- [Background] Sherer DW, Singer G, Uribarri J, Phelps RG, Sapadin AN, Freund KB, Yanuzzi L, Fuchs W, Lebwohl M. Oral phosphate binders in the treatment of pseudoxanthoma elasticum. J Am Acad Dermatol. 2005 Oct;53(4):610-5. doi: 10.1016/j.jaad.2004.11.066. PMID 16198780
- [Background] Blum R, Phelps R, Fuchs W, Lebwohl M. Oral Phosphate Binders in the Treatment of Pseudoxanthoma Elasticum. 64th Annual Meeting American Academy of Dermatology March 3-7, 2006, San Francisco, CA. Manuscript in press J Amer Acad Dermatol 2011
- [Background] Steidl L, Ditmar R. Treatment of soft tissue calcifications with magnesium. Acta Univ Palacki Olomuc Fac Med. 1991;130:273-87. PMID 1838878
- [Background] LaRusso J, Li Q, Jiang Q, Uitto J. Elevated dietary magnesium prevents connective tissue mineralization in a mouse model of pseudoxanthoma elasticum (Abcc6(-/-)). J Invest Dermatol. 2009 Jun;129(6):1388-94. doi: 10.1038/jid.2008.391. Epub 2009 Jan 1. PMID 19122649
- [Background] Iseri LT, French JH. Magnesium: nature's physiologic calcium blocker. Am Heart J. 1984 Jul;108(1):188-93. doi: 10.1016/0002-8703(84)90572-6. No abstract available. PMID 6375330
- [Background] Joffres MR, Reed DM, Yano K. Relationship of magnesium intake and other dietary factors to blood pressure: the Honolulu heart study. Am J Clin Nutr. 1987 Feb;45(2):469-75. doi: 10.1093/ajcn/45.2.469. PMID 3812346
- [Background] Paolisso G, Passariello N, Pizza G, Marrazzo G, Giunta R, Sgambato S, Varricchio M, D'Onofrio F. Dietary magnesium supplements improve B-cell response to glucose and arginine in elderly non-insulin dependent diabetic subjects. Acta Endocrinol (Copenh). 1989 Jul;121(1):16-20. doi: 10.1530/acta.0.1210016. PMID 2662695
- [Background] Rude RK, Singer FR. Magnesium deficiency and excess. Annu Rev Med. 1981;32:245-59. doi: 10.1146/annurev.me.32.020181.001333. No abstract available. PMID 7013665
- [Background] Dietary Reference Intakes for Calcium, Magnesium, Vitamin D and Flouride. IOM Institute of Medicine. 1997 Washington, DC: National Academy Press.
- [Background] Bashir Y, Sneddon JF, Staunton HA, Haywood GA, Simpson IA, McKenna WJ, Camm AJ. Effects of long-term oral magnesium chloride replacement in congestive heart failure secondary to coronary artery disease. Am J Cardiol. 1993 Nov 15;72(15):1156-62. doi: 10.1016/0002-9149(93)90986-m. PMID 8237806
- [Background] Urakabe S, Nakata K, Ando A, Orita Y, Abe H. Hypokalemia and metabolic alkalosis resulting from overuse of magnesium oxide. Jpn Circ J. 1975 Oct;39(10):1135-7. doi: 10.1253/jcj.39.1135. PMID 1195509

RESULTS

PARTICIPANT FLOW:
Groups:
- Magnesium Oxide: Magnesium oxide capsules 800mg twice daily (total of 1000mg of elemental magnesium) for year 1. Upon completion of the first year, barring any safety concerns, all subjects were administered 2500 mg magnesium oxide (total of 1500 mg elemental magnesium) daily for up to one additional year. Subjects received 600 mg elemental magnesium oxide in the morning (taken as two 500 mg magnesium oxide capsules, each containing 300 mg elemental magnesium) and 900 mg elemental magnesium oxide in the evening (taken as three 500 mg magnesium oxide capsules, each containing 300 mg elemental magnesium).
- Placebo: Placebo year 1. Upon completion of the first year, barring any safety concerns, all subjects were administered 2500 mg magnesium oxide (total of 1500 mg elemental magnesium) daily for up to one additional year. Subjects received 600 mg elemental magnesium oxide in the morning (taken as two 500 mg magnesium oxide capsules, each containing 300 mg elemental magnesium) and 900 mg elemental magnesium oxide in the evening (taken as three 500 mg magnesium oxide capsules, each containing 300 mg elemental magnesium).
Period: Placebo-controlled Period
Arm/Group | Magnesium Oxide | Placebo
Started | 22 | 22
Completed | 21 | 20
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2
Period: Open-label Period
Arm/Group | Magnesium Oxide | Placebo
Started | 21 | 20
Completed | 21 | 18
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Magnesium Oxide | Placebo | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.409 (12.764) | 49.364 (12.481) | 49.9 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 18 | 32
  Male | 8 | 4 | 12
Bone Mineral Density (BMD) [Count of Participants; unit: Participants] — Number of participants with low t-score < -1. The T-score is a radiographic diagnosis that compares bone mineral density (BMD) to that of a "normal, healthy, 30-year-old female". The lower the T-score, the lower the BMD. A T-score of +1 to -1 is normal. A T-score decrease of -1 indicates a 10%-15% decrease in BMD.
  Participants
    AP Spine | 3 | 4 | 7
    Forearm | 4 | 4 | 8
    Hip | 1 | 5 | 6
Peau D'Orange right eye [Count of Participants; unit: Participants] — 0 - No evidence of PXE, 1 - Poorly defined, barely visible macules, 2 - Well defined, easily identified macules, 3 - Mostly macules with <5 papules, 4 - >= 5 papules, 5- Patches consisting of confluent macules with <50% of target area covered by papules, 6 - Patches consisting of confluent macules with >=50% of target area covered by papules, 7 - Plaques, 8 - Plaques with mild folds of skin, 9 - Plaques with redundant folds of skin
  Participants
    3 - Mostly macules with <5 papules | 0 | 3 | 3
    4 - >= 5 papules | 22 | 19 | 41
Peau D'Orange left eye [Count of Participants; unit: Participants] — 0 - No evidence of PXE, 1 - Poorly defined, barely visible macules, 2 - Well defined, easily identified macules, 3 - Mostly macules with <5 papules, 4 - >= 5 papules, 5- Patches consisting of confluent macules with <50% of target area covered by papules, 6 - Patches consisting of confluent macules with >=50% of target area covered by papules, 7 - Plaques, 8 - Plaques with mild folds of skin, 9 - Plaques with redundant folds of skin
  Participants
    3 - Mostly macules with <5 papules | 0 | 3 | 3
    4 - >= 5 papules | 22 | 19 | 41
Angioid Streaks right eye [Count of Participants; unit: Participants] — 2- Streaks may be found in association with cardiovascular disease, most commonly of the arterio-sclerotic, hypertensive type 3- Associated with Paget's disease 4- Streaks caused by pigment accumulations and may be termed "secondary"
  Participants
    2 - cardiovascular | 1 | 1 | 2
    3 - Paget's | 0 | 1 | 1
    4 - secondary | 21 | 20 | 41
Angioid Streaks left eye [Count of Participants; unit: Participants]
  2 | 1 | 1 | 2
  3 | 0 | 1 | 1
  4 | 21 | 20 | 41
Subretinal fluid right eye [Count of Participants; unit: Participants]
  N | 20 | 21 | 41
  Y | 2 | 1 | 3
Subretinal fluid left eye [Count of Participants; unit: Participants]
  N | 20 | 20 | 40
  Y | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Von Kossa Staining Per Unit Area of Dermis
Description: A blinded dermatopathologist graded skin biopsies on the density of Von Kossa staining, assessed changes in the amount of calcification of elastic fibers by assessing von Kossa staining per unit area of dermis
Time Frame: up to 2 years
Population: Estimate: Estimated change from baseline and its standard error (SEM). After 1 year=M12-Baseline, After 2 year=M24-Baseline; during 2nd year =M24-M12.
Measure: Mean (Standard Error); unit: microns
Arm/Group | Magnesium Oxide | Placebo
Number analyzed (Participants) | 22 | 22
microns
  After 1 year | -0.0033 (0.0062) | 0.0010 (0.0065)
  during 2nd year | 0.0087 (0.0062) | 0.0123 (0.0070)
  after 2 years | 0.0054 (0.0062) | 0.0132 (0.0069)

2. Secondary Outcome: Number of Participants With a 1-point Decrease of Target Lesions
Description: Changes in skin skin lesions observed through investigator evaluations and clinical photographs. The number of patients with a 1-point decrease of target lesions
Time Frame: up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Magnesium Oxide | Placebo
Number analyzed (Participants) | 22 | 22
Participants
  After 1 year | 2 | 1
  during 2nd year | 8 | 6
  After 2 years | 9 | 7

3. Secondary Outcome: LogMar
Description: Rate of disease progression - Changes observed through ophthalmologic examinations. (+) a decrease in this score indicates improvement of the disease (-) an increase in this score indicates worsening of the disease. LogMAR: logarithm of the minimum angle of resolution. The LogMAR scale converts the geometric sequence of a traditional chart to a linear scale. It measures visual acuity loss: positive values indicate vision loss, while negative values denote normal or better visual acuity.
Time Frame: 2 years
Measure: Mean (Standard Error); unit: LogMar
Arm/Group | Magnesium Oxide | Placebo
Number analyzed (Participants) | 22 | 22
LogMar
  After 1 year | -0.049 (0.036) | -0.063 (0.036)
  during 2nd year | 0.027 (0.041) | 0.015 (0.042)
  After 2 years | -0.022 (0.049) | -0.047 (0.050)

4. Secondary Outcome: VAS - Visual Acuity Score
Description: Rate of disease progression observed through ophthalmologic examinations.(+) an increase in this score indicates improvement of the disease (-) a decrease in this score indicates worsening of the disease. VAS ranges from 10 to 200, with higher score indicating poorer visual acuity.
Time Frame: 2 years
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Magnesium Oxide | Placebo
Number analyzed (Participants) | 22 | 22
units on a scale
  After 1 year | -1.124 (1.141) | -0.602 (1.140)
  during 2nd year | 0.795 (0.927) | -0.729 (0.986)
  After 2 years | -0.329 (1.384) | -1.332 (1.423)

5. Secondary Outcome: Central Retinal Thickness
Description: Rate of disease progression observed through ophthalmologic examinations. (+) a decrease in this scores indicates improvement of the disease; (-) an increase in this scores indicates improvement of the disease.
Time Frame: 2 years
Measure: Mean (Standard Error); unit: µm
Arm/Group | Magnesium Oxide | Placebo
Number analyzed (Participants) | 22 | 22
µm
  After 1 year | 2.965 (0.373) | -3.552 (3.429)
  during 2nd year | -4.203 (3.877) | -6.796 (4.123)
  After 2 years | -1.238 (3.913) | -10.348 (4.143)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Magnesium Oxide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 11/22 | 11/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Magnesium Oxide (N=22) | Placebo (N=22)
Diarrhea (Gastrointestinal disorders) | 10 (14) | 9 (9) — diarrhea
Loose Stool (Gastrointestinal disorders) | 1 (2) | 2 (2)
Abdominal Cramps (Gastrointestinal disorders) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Flatulance (Gastrointestinal disorders) | 0 (0) | 2 (2)
Bloating (Gastrointestinal disorders) | 1 (1) | 1 (1)
Increased bowel movements (Gastrointestinal disorders) | 0 (0) | 2 (2)
Loss of Appetite (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 3 (3)
Upper Respiratory Infection (Infections and infestations) | 0 (0) | 2 (2)
Infections (Infections and infestations) | 1 (1) | 5 (8) — Sinus, Dental, urinary

LIMITATIONS AND CAVEATS:
Small study of a rare disease with tremendous patient variation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes